CLINICAL TRIAL: NCT05542134
Title: Platelet Agregation in Patients on ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Noc, MD PhD, University Medical Centre Ljubljana
Other Study IDs: KOIIM-UM
Record Dates: First submitted 2022-09-01; First posted 2022-09-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Platelet Refractoriness
Keywords: V-A ECMO; platelet reactivity; ECMO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- V-A ECMO without P2Y12 inhibitors: control group
  Interventions: Diagnostic Test: P2Y12 Platelet Aggregation Inhibitor
- V-A ECMO with P2Y12 inhibitor at the time of ECMO: observational group 1
  Interventions: Diagnostic Test: P2Y12 Platelet Aggregation Inhibitor
- V-A ECMO already recieving P2Y12 inhibitors: observational group 2
  Interventions: Diagnostic Test: P2Y12 Platelet Aggregation Inhibitor

INTERVENTIONS:
Diagnostic Test: P2Y12 Platelet Aggregation Inhibitor — Verify now PRU test

SUMMARY:
An observational study in which investigators will observe platelet inhibition in patients on VA ECMO acorrding to treatment with P2Y12 inhibitor.

DETAILED DESCRIPTION:
Investigators will perform an observational study in which platelet inhibition in patients on VA ECMO acorrding to treatment with P2Y12 inhibitor will be observed.

Participants will be divided into three groups:

A: patients on V-A ECMO without P2Y12 inhibitors B patients on V-A ECMO with P2Y12 inhibitors with administration of P2Y12 inhibitor at the time of ECMO insertion C: patients on V-A ECMO already recieving P2Y12 inhibitors at the time of ECMO insertion.

Blood samples will be taken prior to and at 2, 4, 12, 22, 48, 72 after ECMO insertion and after removal of an ECMO. VerifyNow System will be used to measure platelet agregation (PRU test).

ELIGIBILITY:
Inclusion Criteria:

* all patients on VA ECMO

Exclusion Criteria:

* known P2Y12 alergy
* thrombocitopenic patents (< 50*109/L),
* patients treated with eptifibatide ali bivalirudin
* patients younger than 18 years
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patents treated with ECMO.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 2 after VA ECMO insertion)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 4 after VA ECMO insertion)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 12 after VA ECMO insertion)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 22 after VA ECMO insertion)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 48 after VA ECMO insertion)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 72 after VA ECMO insertion)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.
Verify now P2Y12 platelet inhibition | (Time Frame: Hour 24 after VA ECMO removal)
  Platelet inhibition measured by VerifyNow as P2Y12 reaction units (PRU). Platelet reactivity reflects P2Y12 inhibitor effect with higher PRU values showing low P2Y12 response and lower values decreased platelet reactivity due to the effect of a P2Y12 inhibitor.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
If needed we are happy to share data